CLINICAL TRIAL: NCT04014790
Title: An Open Label Phase 2, Study to Evaluate the Safety and Efficacy of RGI-2001 for the Prevention of Acute Graft-vs-Host Disease Compared to Contemporary Controls in Subjects Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: RGI-2001 for the Prevention of Acute Graft-vs-Host Disease in Subjects Following Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RGI-2001-003
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Graft Vs Host Disease; Graft-versus-host-disease; Acute-graft-versus-host Disease; Prevention of aGVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — KRN 7000; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RGI-2001 (Experimental): Subjects will be administered RGI 2001 in combination with standard of care treatment
  Interventions: Drug: RGI-2001; Drug: Standard of Care

INTERVENTIONS:
Drug: RGI-2001 — Subjects will receive 6 weekly doses of RGI 2001, 100 μg/kg via IV administration after completion of alloHSCT
  Other Names: KRN-7000; RGI-7000
Drug: Standard of Care — Standard of care prophylaxis regimen will be administered according to institutional guidelines

SUMMARY:
This Phase II open label study will evaluate the safety and efficacy of repeat doses of RGI-2001 in combination with standard of care treatment for the prevention of acute graft-vs-host-disease (aGvHD) in subjects following Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT). These subjects will be compared to contemporary controls.

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-arm study to evaluate six weekly doses of RGI-2001 in combination with standard of care treatment for the prevention of aGvHD in subjects following alloHSCT. The study will include a Safety Run-in Phase to assess the safety and tolerability of 6 weekly doses of RGI-2001 followed by an Expansion Phase in which the potential efficacy of 6 weekly doses of RGI-2001 in addition to standard of care for GvHD prophylaxis will be assessed. Comparison will be made to a contemporaneous control group.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ≥ 18 and ≤ 65 years of age
2. Has a hematologic malignancy which includes Acute myelogenous leukemia (AML), T or B cell acute lymphoblastic leukemia (ALL) Myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), myeloproliferative disorder (MPD) including myeloid metaplasia and CML
3. Must have adequate organ function
4. Transplant Donor: Matched related donor or Unrelated donor
5. Is a candidate for anti-graft-vs-host-disease (GvHD) prophylaxis that includes a calcineurin inhibitor
6. Ability to understand and willingness to sign a written informed consent form
7. If female of childbearing potential, must have had a negative serum pregnancy test prior to enrollment and must have agreed to use a double barrier method of contraception for 30 days after RGI-2001 administration
8. If male, must be sterile or willing to use an approved method of contraception from the time of informed consent to 90 days after last dose of RGI-2001 administration

Exclusion Criteria:

1. Has had any other prior organ transplantation
2. Planned procedure to deplete regulatory T cells from donor transplant materials
3. Planned reduced intensity conditioning
4. Has had prior treatment with anti-CD3, other T cell depleting antibodies, or anti-thymocyte globulin within 12 months prior to alloHSCT procedure
5. Has progressive underlying malignant disease including post-transplant lymphoproliferative disease
6. Has evidence of active central nervous system (CNS) disease including known brain or leptomeningeal disease (CT or MRI scan of the brain required only in case of clinical suspicion of CNS involvement)
7. Is female and pregnant or lactating
8. Has a documented history of uncontrolled autoimmune disease or on active treatment
9. History of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to receiving study drug

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - UCLA Medical Center, Los Angeles, California
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Irving Medical Center, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeFilipp Z, Choe H, Efebera YA, Saad A, Farhan S, Lekakis L, Yared JA, Schiller G, Mapara MY, Assal A, Gooley T, Bui JD, Lee D, Lane H, Chen YB. RGI-2001 for the prophylaxis of acute graft-versus-host disease after allogeneic HCT. Blood. 2025 Oct 23;146(17):2037-2046. doi: 10.1182/blood.2025029584. PMID 40680268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RGI-2001
Started | 49
Completed | 43
Not Completed | 6
Not completed — Death | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | RGI-2001
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 45
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Grades II-IV aGVHD
Description: Acute GVHD will be graded and assessed according to modified KEYSTONE criteria and the severity grade (Grade II through IV) were captured up through the first 100 days post-transplant
Time Frame: Day 100 post-transplant
Population: intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | RGI-2001
Number analyzed (Participants) | 48
Participants | 11

2. Secondary Outcome: Grades II-IV aGVHD
Description: Acute GVHD will be graded and assessed within 180 days post-transplant
Time Frame: Day 180 post-transplant
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | RGI-2001
Number analyzed (Participants) | 48
Participants | 11

3. Secondary Outcome: Non-relapse Mortality (NRM) Rates
Description: The probability of mortality not preceded by relapse of the underlying malignancy will be estimated
Time Frame: 1 year post-transplant
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | RGI-2001
Number analyzed (Participants) | 48
Participants | 2

4. Secondary Outcome: Disease-free Survival (DFS)
Description: The probability of survival without relapse of the underlying malignancy will be estimated
Time Frame: 1 year post-transplant
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | RGI-2001
Number analyzed (Participants) | 48
Participants | 40

5. Secondary Outcome: GvHD-free, Relapse Free Survival (GRFS)
Description: The probability of survival without relapse of the underlying malignancy, without severe (grades 3-4) acute GVHD, and without chronic GVHD requiring systemic immunosuppression will be estimated
Time Frame: 1 year post-transplant
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | RGI-2001
Number analyzed (Participants) | 48
Participants | 26

6. Secondary Outcome: Overall Survival (OS)
Description: The probability of survival will be estimated
Time Frame: 1 year post-transplant
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | RGI-2001
Number analyzed (Participants) | 48
Participants | 44

ADVERSE EVENTS:
Time Frame: TEAE is defined as any AE reported on or after the first dose date of RGI-2001, or that was already present and worsened after the first dose date, up to 30 days after the last RGI-2001 dose date. TEAE were collected from sign of consent up through 9 weeks after transplant. TEAE for all cause mortality were collected up through 1 year.
Description: TEAE were collected from sign of consent up through 9 weeks after transplant.
Groups:
- RGI-2001: Subjects will be administered RGI 2001 in combination with standard of care treatment (Tacrolimus and Methotrexate)
  RGI-2001: Subjects will receive 6 weekly doses of RGI 2001, 100 μg/kg via IV administration after completion of alloHSCT
  Standard of Care: Standard of care prophylaxis regimen will be administered according to institutional guidelines
Arm/Group | RGI-2001
All-Cause Mortality (participants affected / at risk) | 4/49
Serious Adverse Events (participants affected / at risk) | 8/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGI-2001 (N=49)
Myocarditis (Cardiac disorders) | 1 (1) — Pericarditis
Diarrhea (Gastrointestinal disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) — Sepsis and Acute kidney injury
Headache (Nervous system disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGI-2001 (N=49)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 11 (11)
Stomatitis (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 9 (9)
Fatigue (General disorders) | 7 (7)
Muscosal Inflammation (General disorders) | 6 (6)
Alanine Aminotransferase increased (Investigations) | 6 (6)
Aspartate Aminotransferase increased (Investigations) | 3 (3)
Blood Alkaline Phosphatase Increased (Investigations) | 3 (3)
Blood Creatinine increased (Investigations) | 3 (3)
Blood Lactate Dehyrogenase increased (Investigations) | 3 (3)
Neutrophil Count Decreased (Investigations) | 6 (6)
Platelet Count Decreased (Investigations) | 7 (7)
White blood cell count decreased (Investigations) | 6 (6)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) — maculo-papular, rash papular, rash, rash generalized, rash pruritic, rash follicular
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04014790/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT04014790/SAP_001.pdf